CLINICAL TRIAL: NCT03118102
Title: the Effects of Noise in Operating Rooms on Anesthetists Hearing
Brief Title: Audiological Evaluation of Anesthetists
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, khaled salah mohamed, lecturer of anaesthesia and ICU, Assiut University
Other Study IDs: kmohamed
Record Dates: First submitted 2017-04-09; First posted 2017-04-18 (Actual); Last update posted 2018-01-09 (Actual); Status verified 2018-01

CONDITIONS: Hearing Loss
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- anesthetist group: anesthetist doctor who subjected to noise in operating rooms
- control group: doctors in the same hospital who are not subjected to noise in operating rooms

SUMMARY:
The investigators aim to investigate the effect of operating room noise on anesthetist hearing

ELIGIBILITY:
Inclusion Criteria:

* anesthetist doctor and non-anesthetist doctor less than 40 years

Exclusion Criteria:

* doctors above 40 years

Ages: 28 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: anesthetist doctor who subject to noise in operating rooms
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2017-04-10 (Actual); Primary Completion 2018-01-08 (Actual); Study Completion 2018-01-08 (Actual)

PRIMARY OUTCOMES:
Extended high frequency audiometry | 20 minutes
  pure tone audiometry in the frequency range from 250Hz-20,000Hz

SECONDARY OUTCOMES:
Transient Evoked Otoacoustic Emission | 10 minutes
  stimulus induced cochlear echos in the frequency range from 1000-4000 Hz

CONTACTS AND LOCATIONS:
Overall Officials: Khaled Salah Mohamed, MD, Principal Investigator — Assiut University
Locations (1):
- Assiut university hospital, Asyut, Egypt